CLINICAL TRIAL: NCT06640959
Title: Chronic Radiation Induced Bowel Toxicity Study (CRIBS)
Brief Title: Chronic Radiation Induced Bowel Toxicity Study
Acronym: CRIBS
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other); Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTsp225
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, blood samples, mid-stream urine samples, optional rectal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Procedure - blood, urine and stool sample collection — Samples will be collected (blood, urine, stool and optional rectal swab) at baseline (prior to the start of radiotherapy), weekly during radiotherapy for 4 weeks, 6-8 weeks and 12 weeks from start of radiotherapy, and at 6-month and 12-month follow-up appointments

SUMMARY:
In the UK over 22,000 people undergo pelvic radiotherapy treatment per year, for several types of cancers including prostate cancer. The investigators want to investigate whether there are any differences in the bacteria in the bowel in patients with prostate cancer and whether these change during treatment.

The aim of this study is to analyse the bacteria from the stool of patients undergoing radiotherapy for prostate cancer. The investigators will also look for any changes in the urine, blood and using rectal swabs that might be a surrogate for what is happening in the gut at the same time. They will collect food frequency/ food diary information for each patient alongside health questionnaires.

The investigators aim to recruit approximately 50 patients diagnosed with prostate cancer due to undergo radiotherapy over a two year period. Patients will be recruited across 2 sites (Rosemere Cancer Centre, Lancashire Teaching Hospitals Trust and The Christie NHS Foundation Trust).

DETAILED DESCRIPTION:
This is a prospective, translational study which aims to investigate the radiation induced immunological changes in the bowel mucosa, blood and urine, and the role of the microbiota in acute and late bowel toxicity.

The investigators aim to recruit 50 patients newly diagnosed with (histologically confirmed) localised, intermediate to high-risk prostate cancer (T2b -T4a N0 M0), who are due to undergo standard of care radical radiotherapy (Intensity modulated radiotherapy (IMRT)) (60Gy in 20# with curative intent) 4-week regimen.

Eligible patients who have consented to the study will provide the following samples at baseline (prior to the start of radiotherapy), weekly during radiotherapy for 4 weeks, 6-8 weeks and 12 from the start of radiotherapy, and at 6-month and 12-month follow-up appointments:

1. stool sample
2. blood sample (40mls) delegated nurse or research nurse.
3. mid-stream urine sample
4. optional rectal swab
5. quality of life health questionnaire

4-day diet diaries will be completed by the patients in the 4 days prior to providing their baseline stool samples and at follow-up appointments (6-8 weeks, 6 months, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥ 18; no upper age limit and able to give informed consent.
* Newly diagnosed patients with, histologically confirmed, localised, intermediate to high-risk prostate cancer (T2b -T4a N0 M0).
* Patients to be treated with prostate radical radiotherapy IMRT (60Gy in 20# with curative intent) 4-week regimen.
* Performance status - ECOG 0-2.

Exclusion Criteria:

* Had received systemic antibiotics (intravenous, intramuscular, or oral) within 2 months before enrolment.
* Had received cytotoxic or immunosuppressive therapies within 6 months of enrolment, including chemotherapy or immunotherapy.
* Had consumed large doses of commercial probiotics (greater or equal to 108 CFU per day) within 12 months of enrolment (such as Actimint®, CranProBio®, ImmunoProBio®, among others).
* Patients with diagnosed inflammatory bowel disease or coeliac disease
* Patients with previous colorectal cancer
* Patients who have undergone colectomy (total or subtotal)
* Patients with a history of diverticulitis (uncomplicated diverticular disease permitted)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of obtaining longitudinal blood, urine and stool samples | From enrolment until 12 months post treatment
  Feasibility of obtaining longitudinal blood, urine and stool samples from patients with newly diagnosed prostate cancer undergoing standard of care radiotherapy.
  Samples will be collected at baseline (prior to the start of radiotherapy), weekly during radiotherapy for 4 weeks, 6-8 weeks and 12 from the start of radiotherapy, and at 6-month and 12-month follow-up appointments.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston, Lancashire

IPD SHARING:
Plan to Share IPD: No